CLINICAL TRIAL: NCT03099265
Title: Phase II Study to Evaluate Neoadjuvant Modified FOLFIRINOX and Stereotactic Body Radiation Therapy in Borderline Resectable Pancreatic Adenocarcinoma
Brief Title: Neoadjuvant Modified FOLFIRINOX and Stereotactic Body Radiation Therapy in Borderline Resectable Pancreatic Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Paused due to COVID. A determination was made to stop the study because it would be impossible to reach the 65% resection rate as outlined in the protocol.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000020432
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Results first posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- patients with borderline resectable pancreatic adenocarcinoma (Experimental): Borderline resectable disease will be defined by NCCN criteria, and determined centrally by review of a diagnostic pancreas protocol CT scan and/or MRI scan with contrast by a dedicated surgical oncologist and radiologist.
  Interventions: Drug: neoadjuvant mFOLFIRINOX; Drug: Stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Drug: neoadjuvant mFOLFIRINOX — Patients will receive 8 cycles of mFOLFIRINOX every 2 weeks. mFOLFIRINOX will be dosed as follows: Oxaliplatin 85 mg/m2, followed by folinic acid 400 mg/m2 infused over 120 minutes and irinotecan 135 mg/m2 infused over 90 minutes, followed by 5-fluorouracil 300 mg/m2 IV bolus, followed by 2,400 mg/m2 continuous infusion for 46 hours. Levoleucovorin may be substituted for folinic acid at a dose of 200 mg/m2 infused over 120 minutes.
  Other Names: Oxaliplatin; Irinotecan; Leucovorin; 5-fluorouracil; folinic acid
Drug: Stereotactic body radiotherapy (SBRT) — Stereotactic body radiotherapy (SBRT) will be delivered to the primary tumor and any adjacent involved nodes to 33 Gy in 5 fractions over the course of 2 weeks, and within 4 weeks of chemotherapy.

SUMMARY:
Surgical resection is the only potentially curative treatment for patients with pancreatic cancer. Patients with BRPC have tumors in close contact with the vasculature but not to the extent that resection is prohibited. Nonetheless, retrospective studies have shown that immediate resection in these patients is associated with an increased risk of positive margins, and a margin positive resection does not improve survival over that of patients with unresectable disease. Moreover, even in those patients where a successful resection is achieved, there is a high rate of early metastatic progression suggesting that micrometastatic disease is often present at diagnosis. Therefore neoadjuvant therapy is likely to improve outcomes in patients with BRPC to increase the likelihood of achieving a margin negative resection, provide early control of occult micrometastatic disease, and select those patients without systemic progression who would benefit from surgical resection.

DETAILED DESCRIPTION:
Given the superior outcomes with FOLFIRINOX and the potential for improved local response with SBRT, the investigators propose to evaluate the efficacy of pre-operative modified FOLFIRINOX followed by SBRT in patients with borderline resectable pancreatic adenocarcinoma. The investigators hypothesize that pre-operative modified FOLFIRINOX followed by SBRT will improve the rate of R0 resections compared to historical controls treated with standard gemcitabine-based chemotherapy and fractionated radiation prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed pancreatic adenocarcinoma
* Borderline resectable pancreatic adenocarcinoma, determined centrally by review of a diagnostic CT scan and/or MRI scan with contrast by a dedicated surgical oncologist and radiologist, or as determined by EUS, and defined according to the NCCN consensus guidelines
* ECOG Performance Status of 0-1
* Age > 18
* Laboratory parameters as follows:

  * Absolute neutrophil count >=1,500/uL
  * Platelet count >=100,000/uL
  * Hemoglobin >=9 g/dL
  * Creatinine <1.5 X ULN or estimated GFR >30 ml/min
  * Bilirubin =<1.5 X ULN
  * AST and ALT =<3 X ULN
  * Negative pregnancy test in women of childbearing potential
* Able to have fiducials placed in the pancreas
* Patients who received chemotherapy >5 years ago for malignancies other than pancreatic cancer are eligible

Exclusion Criteria:

* Evidence of extrapancreatic disease on diagnostic imaging (CT, MRI, or PET scan), or laparoscopy, including nodal involvement beyond the peripancreatic tissues and/or distant metastases
* Evidence of invasion into the duodenum or stomach, as determined by EGD/EUS
* Prior treatment (chemotherapy, biological therapy, or radiotherapy) for pancreatic cancer
* Prior treatment with oxaliplatin, irinotecan, fluoruouracil or capecitabine
* Major surgery within 4 weeks of study entry
* Other concurrent anticancer therapies
* Other malignancy within the past five years (exceptions include basal cell carcinoma of the skin, cervical carcinoma in situ, and non-metastatic prostate cancer)
* Evidence of second malignancy at the time of study entry
* Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* Grade 2 or greater sensory peripheral neuropathy
* Uncontrolled seizure disorder, active neurological disease, or known CNS disease
* Significant cardiac disease, including the following: unstable angina, New York Heart Association class II-IV congestive heart failure, myocardial infarction within six months prior to study enrollment
* Pregnant or nursing
* Other medical condition or reason that, in the opinion of the investigator, would preclude study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Johung, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Smilow Cancer Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Borderline Resectable Pancreatic Adenocarcinoma
Started | 9
Per Protocol Week 12 | 8
Per Protocol Week 24 | 4
Completed | 8
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Of 11 patients, 9 were eligible to be enrolled.
Arm/Group | Patients With Borderline Resectable Pancreatic Adenocarcinoma
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With and Without R0 Resection
Description: The primary outcome of this study is the R0 resection count of patients with BRPC treated with neoadjuvant mFOLFIRINOX and SBRT. R0 resection indicates a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed. When the study results were entered, rate was replaced with count as the manner in which these data were summarized.
Time Frame: Up to 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Borderline Resectable Pancreatic Adenocarcinoma
Number analyzed (Participants) | 9
Participants
  Yes | 2
  No | 7

2. Secondary Outcome: Number of Participants Response to Neoadjuvant Therapy Using RECIST
Description: Response to treatment will be assessed by the treating physicians and investigators according to RECIST version 1.1. Counts of participants' RECIST category at their final visit up to 40 weeks below are provided. Per Response Evaluation Criteria In Solid TumorsCriteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response(CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Borderline Resectable Pancreatic Adenocarcinoma
Number analyzed (Participants) | 9
Participants
  stable disease (SD) | 7
  progressive disease (PD) | 1
  partial response (PR) | 1

3. Secondary Outcome: Number of Participants With and Without Pathologic Response to Neoadjuvant Therapy
Description: A pathologic complete response is defined as the absence of residual invasive disease at the completion of the neoadjuvant treatment. This was performed only in those that had R0 resection performed.
Time Frame: Up to 40 weeks
Population: Only patients with R0 resection had pathologic response assesssed.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Borderline Resectable Pancreatic Adenocarcinoma
Number analyzed (Participants) | 2
Participants
  Yes | 0
  No | 2

4. Secondary Outcome: Number of Participants With and Without Recurrence
Description: Number of participants with and without recurrence following surgery. This outcome was updated when the results were entered.
Time Frame: Up to 40 weeks
Population: This population includes the 8 of 9 patients that experienced disease progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Borderline Resectable Pancreatic Adenocarcinoma
Number analyzed (Participants) | 8
Participants
  Local Progression | 4
  Metastatic Progression | 4

5. Secondary Outcome: Number of Participants: Progression Free Survival
Description: Presented are count of patients that had experienced either progression free survival or disease progression through the follow up period.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Borderline Resectable Pancreatic Adenocarcinoma
Number analyzed (Participants) | 9
Participants
  Progression Free Survival | 1
  Disease Progression | 8

6. Secondary Outcome: Number of Participants: Overall Survival
Description: Presented are counts of patients that we either deceased or not deceased at the end of the follow up period.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Borderline Resectable Pancreatic Adenocarcinoma
Number analyzed (Participants) | 9
Participants
  Deceased | 6
  Not Deceased | 3

7. Secondary Outcome: Grade 3 or Greater Acute and Late Gastrointestinal Toxicity
Description: To determine rates of grade 3 or greater gastrointestinal toxicity, including acute toxicities occurring within 3 months of treatment, and late toxicities occurring over 3 months after completion of radiation. This outcome was clarified when results were entered. The number of patients that experienced at least 1 grade 3 (or greater) event are presented.
Time Frame: Up to 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Borderline Resectable Pancreatic Adenocarcinoma
Number analyzed (Participants) | 9
Participants | 5

ADVERSE EVENTS:
Time Frame: Up to 40 weeks
Arm/Group | Patients With Borderline Resectable Pancreatic Adenocarcinoma
All-Cause Mortality (participants affected / at risk) | 6/9
Serious Adverse Events (participants affected / at risk) | 6/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Borderline Resectable Pancreatic Adenocarcinoma (N=9)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Hepatobility disorders - Other, specify (Hepatobiliary disorders) | 1 (1) — Jaundice/ Elevated bilirubin
Sepsis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Borderline Resectable Pancreatic Adenocarcinoma (N=9)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (5)
Infections and infestations - Other, specify (Infections and infestations) | 2 (3)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (2)
Alanine aminotransferase increased (Investigations) | 3 (5)
Alkaline phosphatase increased (Investigations) | 3 (6)
Aspartate aminotransferase increased (Investigations) | 2 (6)
Blood bilirubin increased (Investigations) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (2)
Weight loss (Investigations) | 5 (11)
White blood cell decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 8 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Amnesia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (4)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (7)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 6 (6)
Palpitations (Cardiac disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (2)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (9)
Constipation (Gastrointestinal disorders) | 7 (9)
Diarrhea (Gastrointestinal disorders) | 7 (19)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4 (5)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (12)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (4)
Oral dysesthesia (Gastrointestinal disorders) | 2 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 (6)
Fatigue (General disorders) | 9 (16)
Gait disturbance (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 6 (10)
Irritability (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Edema limbs (General disorders) | 3 (3)
Infusion related reaction (General disorders) | 4 (4)
Non-cardiac chest pain (General disorders) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT03099265/Prot_SAP_000.pdf